CLINICAL TRIAL: NCT03819218
Title: A Multicentre, Open-label, Single-group Maximal Use Trial, Evaluating the Safety and Pharmacokinetic Profile of the Active Ingredients and Their Metabolites After Application of MC2-01 Cream in Adolescents With Extensive Psoriasis Vulgaris
Brief Title: A Maximal Use Trial Evaluating the Pharmacokinetic Profile of MC2-01 Cream in Adolescent Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: MC2 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC2-01-C6
Record Dates: First submitted 2019-01-11; First posted 2019-01-28 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-02

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MC2-01 cream (Experimental): MC2-01 (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream. One application daily for 8 weeks
  Interventions: Drug: MC2-01 cream

INTERVENTIONS:
Drug: MC2-01 cream — MC2-01 cream (Calcipotriene/betamethasone dipropionate, w/w 0.005%/ 0.064%)

SUMMARY:
This is a phase 2, open-label, single-group, multicentre trial in which the investigational product, MC2-01 cream, is investigated in adolescent subjects (age 12 to 16 years, 11 months) with clinically diagnosed extensive psoriasis vulgaris.

DETAILED DESCRIPTION:
The MC2-01 cream is designed for optimal patient satisfaction - it quickly absorbs into the skin leaving it nicely moisturized allowing patients to move on with daily routines. In this trial, subjects who fulfil all inclusion and exclusion criteria are enrolled in the trial and will apply one dose of trial medication topically once daily for 8 weeks. The purpose of the trial, is to determine the and pharmacokinetic parameters of MC2-01 cream in adolescent subjects under maximum use conditions.

ELIGIBILITY:
Inclusion Criteria:

* The parent(s), or legal guardian(s) (according to national law) have provided written informed consent following their receipt of verbal and written information about the trial
* The subject (according to national law) has provided written assent to the trial following their receipt of verbal and written information about the trial
* Generally healthy males or non-pregnant females, of any race or ethnicity, who are between 12 to 16 years, 11-month-old at Screening Visit 1 (SV1)
* At Visit 1/Day 0, have a clinical diagnosis of plaque psoriasis (psoriasis vulgaris) of at least 6 months duration involving body (trunk and/or limbs), with or without scalp
* Have a treatment area between 10% and 30% of the Body Surface Area (BSA) on the body (trunk and/or limbs) and scalp, excluding psoriatic lesions on the face, genitals, and intertriginous areas, at Visit 1/Day 0
* Have a Physician's Global Assessment (PGA) of at least moderate severity on the treatment area
* A normal HPA axis function including a serum cortisol concentration above 4,5 mcg/dl before ACTH-challenge and equal or above 18 mcg/dl 30 minutes after ACTH challenge, at Screening Visit 2 (SV2)
* A serum albumin-corrected calcium below the upper reference limit at SV2

Exclusion Criteria:

* Have a current diagnosis of unstable forms of psoriasis, including erythrodermic or pustular psoriasis
* Other inflammatory skin disease in the treatment area that may confound the evaluation of the psoriasis vulgaris
* Presence of infections in the treatment area or skin manifestations or atrophic skin, atrophic striae, skin vein fragility, ichthyosis, acne vulgaris, acne rosacea, rosacea, ulcers and wounds in the treatment area
* Presence of pigmentation, extensive scarring, pigmented lesions or sunburn in the treatment areas, which could interfere with the rating of efficacy parameters
* Planned excessive or prolonged exposure to either natural or artificial sunlight
* Use of phototherapy (psoralen + ultraviolet A radiation and ultraviolet B radiation within 4 weeks prior to SV2 and during the trial
* Current or past history of disorders of calcium metabolism associated with hypercalcemia, vitamin D toxicity, severe renal insufficiency, or severe hepatic disorders
* Oral calcium supplements, vitamin D supplements, bisphosphonates or calcitonin within 4 weeks prior to SV2
* Planned initiation of, or changes to concomitant medication that could affect calcium metabolism during the trial;
* Planned initiation of, or changes to, concomitant estrogen therapy during the trial
* Strong systemic cytochrome P450 3A4 (CYP 3A4) inhibitors or inducers within 4 weeks prior to SV2 and during the trial
* Use of topical treatments, except for emollients and non-medicated shampoos, with a possible effect on psoriasis within 2 weeks prior to SV2 and during the trial
* Systemic treatment with biological therapies, with a possible effect on psoriasis vulgaris within the following time period prior to SV2 and during the trial
* Initiation of, or expected changes to, concomitant medication that may affect psoriasis during the trial
* Any of the following conditions, whether known or suspected; Clinically diagnosed depression where the subject is in current treatment with medication approved for treatment of depression; Endocrine disorders known to affect cortisol levels or HPA axis integrity; Non-nocturnal sleep patterns
* Use of systemic medication that suppresses the immune system and other systemic chemotherapeutic antineoplastic therapy within 4 weeks prior to the SV2 and during the trial
* Use of live vaccines 4 weeks before SV2 and during the trial
* Have clinical signs of skin infection with bacteria, viruses, or fungi
* Known human immunodeficiency virus (HIV) infection, active hepatitis B or hepatitis C
* Known or suspected of hypersensitivity to any component of the test product
* Known allergic asthma, serious allergies or allergies where recurrent acute or chronic treatment is necessary
* Have any chronic or acute medical condition that, in the opinion of the investigator, may pose a risk to the safety of the subject, or may interfere with the assessment of safety or efficacy in this trial
* Require the use of any concomitant medication that, in the investigator's opinion, has the potential to cause an adverse effect when given with the Investigational Product (IP) or will interfere with the interpretation of the trial results
* Subject with known abnormal reduction in muscle mass, as judged by the investigator

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Pinter, MD, Principal Investigator — Dept. of Dermatology, Venereology and Allergology
Locations (2):
- PRO SANUM a.s., Prague, Czechia
- Dept. of Dermatology, Venereology and Allergology, Frankfurt, Frankfurt/Main, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MC2-01 Cream
Started | 7
Completed | 6
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Czechia | 5
  Germany | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HPA (Hypothalamic-pituitary-adrenal) Axis Suppression at Week 4
Description: Adrenal function will be assessed in a challenge test with an intravenous dose of cosyntropin. Measurement of serum cortisol levels pre- and post- stimulation is an accepted standard method used to evaluate adrenal suppression.
  The test consists of an initial blood sampling. Following the blood sample, an intravenous bolus injection of 0.25 mg cosyntropin is given. The serum cortisol concentration 30 min. after will reflect stimulation of the adrenal glands induced by cosyntropin. HPA axis suppression is define as serum cortisol below 18 µg/dL
Time Frame: Week 4
Population: The HPA population was defined as all subjects in the safety population that showed a normal HPA function at the screening visit.
Measure: Count of Participants; unit: Participants
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Number of Participants With HPA (Hypothalamic-pituitary-adrenal) Axis Suppression at Week 8
Description: as for outcome 1
Time Frame: Week 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 6
Participants | 0

3. Primary Outcome: Change in S-Calcium Metabolism at Week 4
Description: Change from Baseline to Week 4 in albumin-corrected S-calcium
Time Frame: Week 4
Population: 7 subjects were included in the safety population at baseline and Week 4. At Week 8 1 subjects was withdrawn.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 7
mmol/L | -0.037 (0.084)

4. Primary Outcome: Change in S-Calcium Metabolism at Week 8
Description: Change from Baseline to Week 8 in albumin-corrected S-calcium
Time Frame: Week 8
Population: 7 subjects were included in the safety population at baseline and Week 4. At Week 8 1 subjects was withdrawn.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 7
mmol/L | -0.027 (0.060)

5. Primary Outcome: Change in U-Calcium Metabolism at Week 4
Description: Change from Baseline to Week 4 in Urinary Calcium/Creatinine ratio (mol/mol)
Time Frame: Week 4
Population: 7 subjects were included in the safety population at baseline and Week 4. At Week 8 1 subjects was withdrawn.
Measure: Mean (Standard Deviation); unit: mol/mol
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 7
mol/mol | 0.115 (0.426)

6. Primary Outcome: Change in U-Calcium Metabolism at Week 8
Description: Change from Baseline to Week 8 in Urinary Calcium/Creatinine ratio (mol/mol)
Time Frame: Week 8
Population: 7 subjects were included in the safety population at baseline and Week 4. At Week 8 1 subjects was withdrawn.
Measure: Mean (Standard Deviation); unit: mol/mol
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 7
mol/mol | 0.058 (0,186)

7. Secondary Outcome: The Maximum Plasma Concentration [Cmax] of Betamethasone 17-propionate at Week 4
Description: The Maximum Plasma Concentration [Cmax] of the metabolite of BDP, betamethasone 17-propionate measured at Week 4.
Time Frame: Week 4
Population: The Maximum Plasma Concentration [Cmax] of the metabolite of BDP, betamethasone 17-propionate, was quantifiable in 3 out of 6 (50 %) participants only, thus the data only reflects result from 3 participants. The 3 remaining participants had values below Lower Limit of Quantification (LLOQ).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 6
pg/mL | 37.53 (22.82)

8. Secondary Outcome: Time to Maximum Plasma Drug Concentration [Tmax] of Betamethasone 17-propionate at Week 4
Description: Time to maximum plasma drug concentration [Tmax] of the metabolite of BDP, betamethasone 17-propionate measured at Week 4.
Time Frame: Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | MC2-01 Cream
Number analyzed (Participants) | 6
Hours | 2.333 (1.155)

ADVERSE EVENTS:
Time Frame: AEs were collected/assessed from the time of the signature of the informed consent form by the participant and until the final follow-up visit has occurred, i.e. up to in total up to 18 weeks, including a screening period of up to 6 weeks, a treatment period of 8 weeks and a follow-up period of 4 weeks. AEs that were considered related to the trial product would be followed until they were resolved, or until the medical condition of the participant was stable.
Arm/Group | MC2-01 Cream
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MC2-01 Cream (N=7)
Nasopharyngitis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-09-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT03819218/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT03819218/SAP_001.pdf